CLINICAL TRIAL: NCT03891134
Title: Associated Risk Factors and Effect of Nutritional Intervention for Sarcopenia and Constipation in Middle-Aged and Old People
Brief Title: Nutritional Intervention for Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chimei Medical Center (Other)
Collaborators: The Taiwanese Osteoporosis Association. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMMC10504-J01
Record Dates: First submitted 2019-03-03; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2016-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Amino Acids, Branched-Chain

STUDY DESIGN:
Intervention Model Description: quasi-experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- enriched Branched Chain Amino Acid intervention (Experimental): enriched Branched Chain Amino Acid nutrition supplement 3.6 g twice a day for 5 weeks then withdrawal nutrition supplement for 12 weeks
  Interventions: Dietary Supplement: Branched Chain Amino Acid

INTERVENTIONS:
Dietary Supplement: Branched Chain Amino Acid — Participants were purposively sampled to receive one sachet enriched BCAA twice a day(7.2g) for 5 weeks.

SUMMARY:
Sarcopenia is an age-related poor healthy outcome. nutrition intervention is one , progressive, generalized loss of muscle mass and the decrement in physical activity. Sarcopenia is associated with subsequent health hazards such as disability, falls, functional degeneration, hospitalization and death. There are similar causes between sarcopenia and constipation such as aging, reduced mobility, changes in diet and co-morbidities. Nutrition plays an important role for muscle maintenance. The trial tries to figure out the effect of enriched branched-chain amino acid (BCAA) nutrient on muscle mass, strength and physical performance of sarcopenia in the middle-aged and old people.

DETAILED DESCRIPTION:
Sarcopenia is the progressive loss of skeletal muscle that comes with aging. The population in the World Health Organization (WHO) is ageing rapidly and the proportion of people aged 65 and older will get forecast to increase 25% in 2050. In aging society, sarcopenia has been valued in countries all over the world. The appearance of sarcopenia is associated with decreased physical function, falls, fractures, disability, hospitalization, and poor quality of life. Constipation is a common healthy problem. Similar mechanism and risk factors between sarcopenia and constipation are observed with the association of nutrition, but the interrelationships between them is rarely studied.

Prevention and treatment of sarcopenia is more and more important in the health care. Exercise has positive effects in muscle mass and strength but frail elder can't perform exactly. In addition, dietary intervention is one of the major key to reduce the rate of muscle mass loss and maintain physical performance and function.

Recent studies have found that daily and/or supplemental protein is effective prevention of sarcopenia. Protein is composed of amino acids that can induce a muscle protein anabolic response conditioned by the availability of branched-chain amino acids (such as leucine, isoleucine, valine). Delayed amino acid absorption and anabolic resistance are frequently noted among elderly. Branched chain amino acid (BCAA) or leucine supplementation stimulates muscle protein synthesis.

The recommendation about nutrition for preventing sarcopenia was still inconsistent. The time of study for muscle parameter improvement varies from three days to seven days. At present, there is no consensus about the optimal type of nutritional supplements and hint of how long does nutrition take.

The aim of the present study is to evaluate the influence of enriched BCAA on those people with pre-sarcopenia or sarcopenia. The hypothesis is that subjects after enriched-BCAA supplement improves their physical function, muscle strength, and muscle mass. Subsequently, when dis-continued enriched-BCAA muscle-related outcomes would decline.

ELIGIBILITY:
Inclusion Criteria:

* over 40 years of age
* generally healthy according to responses to a standard health-screening questionnaire.

Exclusion Criteria:

* uncontrolled hypertension or diabetes
* stroke
* severe liver or renal disease
* gastrointestinal disease
* neuromuscular disease
* infectious disease
* cancer,
* pulmonary disease
* disease of the endocrine system
* history of seizures, neurological or significant psychiatric illness
* sensitivity to study ingredients.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle mass index | 0 week
  Skeletal muscle mass index was measured by bioelectrical impedance analysis (BC-418, Tanita)
Skeletal muscle mass index | 5 weeks
  Skeletal muscle mass index was measured by bioelectrical impedance analysis (BC-418, Tanita)
Skeletal muscle mass index | 17 weeks
  Skeletal muscle mass index was measured by bioelectrical impedance analysis (BC-418, Tanita)
Handgrip | 0 weeks
  Grip strength was measured by Grip-D; TKK 5401
Handgrip | 5 weeks
  Grip strength was measured by Grip-D; TKK 5401
Handgrip | 17 weeks
  Grip strength was measured by Grip-D; TKK 5401
6-meter gait speed | 0 weeks
  Measure walking speed of six meters
6-meter gait speed | 5 weeks
  Measure walking speed of six meters
6-meter gait speed | 17 weeks
  Measure walking speed of six meters

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Janssen I, Heymsfield SB, Ross R. Low relative skeletal muscle mass (sarcopenia) in older persons is associated with functional impairment and physical disability. J Am Geriatr Soc. 2002 May;50(5):889-96. doi: 10.1046/j.1532-5415.2002.50216.x. PMID 12028177